CLINICAL TRIAL: NCT02940756
Title: Efficacy and Safety of Artesunate-amodiaquine, Artemether-lumefantrine and Dihydroartemisinine-piperaquine in the Treatment of Uncomplicated Plasmodium Falciparum Malaria in the Democratic Republic of Congo: a Randomized Controlled Trial
Brief Title: Efficacy and Safety of Artemisinin-based Combination Treatments in the Democratic Republic of the Congo
Acronym: TETRDC2016
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ministry of Public Health, Democratic Republic of the Congo (Other Government)
Responsible Party: Principal Investigator, Prof. Gauthier Mesia Kahunu, Professor, Ministry of Public Health, Democratic Republic of the Congo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASAQ-LA-DHAPQP 2015 DRC
Record Dates: First submitted 2016-10-19; First posted 2016-10-21 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-11

CONDITIONS: Malaria
Keywords: Malaria, efficacy, safety, ACT, DR Congo
MeSH Terms: conditions — Malaria | interventions — amodiaquine, artesunate drug combination; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- artesunate-amodiaquine (Experimental): Tablets containing 25 mg of artesunate and 67.5 mg of amodiaquine: one tablet daily for three days children weighing 4.5 to 8 kg, and tablets containing 50 mg of artesunate and 135 mg of amodiaquine: one tablet daily for three days for children weighing 9 to 17 kg.
  Interventions: Drug: artesunate-amodiaquine
- artemether-lumefantrine (Experimental): Tablets containing 20 mg of Artemether and 120 mg of Lumefantrine. Each dose to be taken with high-fat food or drinks (for example milk).
  One tablet twice daily for children weighing 5 to <15 kg, two tablets twice daily for those weighing 15 to <25 kg and three tablets twice daily for those weighing 25 to < 35 kg, for three days.
  Interventions: Drug: artemether-lumefantrine
- Dihydroartemisinine-piperaquine (Experimental): Tablets containing 20 mg of dihydroartemisinine and 160 mg of piperaquine. Half a tablet once daily for children weighing 5 to <7 kg, one tablet once daily for those weighing 7 to <13 kg, and two tablets once daily for those weighing 13 to <24 kg, for three days.
  Interventions: Drug: Dihydroartemisinine-piperaquine

INTERVENTIONS:
Drug: artesunate-amodiaquine — Tablets containing 25 mg of artesunate and 67.5 mg of amodiaquine: one tablet daily for three days children weighing 4.5 to 8 kg, and tablets containing 50 mg of artesunate and 135 mg of amodiaquine: one tablet daily for three days for children weighing 9 to 17 kg.
  Other Names: artesunate-amodiaquine Winthrop®
  Arms: artesunate-amodiaquine
Drug: artemether-lumefantrine — Tablets containing 20 mg of Artemether and 120 mg of Lumefantrine. Each dose to be taken with high-fat food or drinks (for example milk).
  One tablet twice daily for children weighing 5 to <15 kg, two tablets twice daily for those weighing 15 to <25 kg and three tablets twice daily for those weighing 25 to < 35 kg, for three days.
  Other Names: Coartem®
  Arms: artemether-lumefantrine
Drug: Dihydroartemisinine-piperaquine — Tablets containing 20 mg of dihydroartemisinine and 160 mg of piperaquine. Half a tablet once daily for children weighing 5 to <7 kg, one tablet once daily for those weighing 7 to <13 kg, and two tablets once daily for those weighing 13 to <24 kg, for three days.
  Other Names: Eurartesim®
  Arms: Dihydroartemisinine-piperaquine

SUMMARY:
The Democratic Republic of the Congo (DRC) is among the countries most affected by malaria in Sub-Saharan Africa. Condidering its size and the geographic position, the DRC is meant to play a major role in the malaria control in the region. The National Malaria Control program recommends artemisinin-based combination treatments (ACTs), in particular artesunate-amodiaquine or artemether-lumefrantrine for the treatment of uncomplicated malaria. Previous studies indicated that ACTs are still effective, with efficacy above the required threshold of 90%. It is required to assess regularly the efficacy of antimalarial drugs, in order to ascertain the relevance of treatment guidelines such that, in case of increasing failure rates, alternative options can be decided ontime.

The purpose of this trial is to assess efficacy and safety of artesunate-amodiaquine (ASAQ Winthrop®), artemether-lumefantrine (Coartem Dispersible®) and dihydro-artemisinin-piperaquine (Eurartesim®) at day 42 in the treatment of uncomplicated Plasmodium falciparum malaria in six surveillance sites around DRC.

DETAILED DESCRIPTION:
This is a phase 4, randomized, open labelled clinical trial, aiming to assess efficacy and safety of 3 ACTs in the treatment of uncomplicated malaria in the Democratic Republic of the Congo. Children diagnosed with uncomplicated Plasmodium falciparum uncomplicated malaria will be randomized and followed-up during 42 days.

ELIGIBILITY:
Inclusion Criteria:

* children aged 6 to 59 months
* axillary temperature ≥ 37.5 °C or history of fever during the 24 h before recruitment
* monoinfection with Plasmodium falciparum with asexual parasite count of 2,000 to 200,000/µL
* ability to swallow oral medication
* ability and willingness to comply with the protocol for the duration of the study and to comply with the study visit schedule
* informed consent from a parent/guardian
* absence of general danger signs or signs of severe falciparum malaria according to the definitions of WHO (2000)
* absence of severe malnutrition according to WHO child growth standards
* absence of febrile condition due to diseases other than malaria (e.g. measles, acute lower respiratory tract infection, severe diarrhoea with dehydration) or other known underlying chronic or severe diseases (e.g. cardiac, renal or hepatic diseases, HIV/AIDS)
* absence of regular medication, which might interfere with antimalarial pharmacokinetics
* absence of history of hypersensitivity reactions or contraindication to any medicine being tested or used as alternative treatment

Exclusion Criteria:

* presence of general danger signs in children aged under 5 years or signs of severe falciparum malaria according to the definitions of WHO
* body weight < 5kg
* hemoglobin level < 5g/ dL
* mixed or monoinfection with another Plasmodium species detected by microscopy
* presence of severe malnutrition
* presence of febrile conditions due to diseases other than malaria (e.g. measles, acute lower respiratory tract infection, severe diarrhoea with dehydration) or other known underlying chronic or severe diseases (e.g. cardiac, renal and hepatic diseases, HIV/AIDS)
* regular medication, which may interfere with antimalarial pharmacokinetics;
* history of hypersensitivity reactions or contraindications to any of the medicine(s) being tested or used as alternative treatment(s)

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1615 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2018-01-02 (Actual); Study Completion 2018-01-02 (Actual)

PRIMARY OUTCOMES:
PCR-adjusted efficacy | day 42
  the proportion of children with PCR adequate clinical and parasitological response

SECONDARY OUTCOMES:
PCR-unadjusted efficacy | day 42
  the proportion of children with treatment failure: all treatment failures detected during the follow-up, regardless of genotyping
K-13 propeller polymorphisms | day 42
  the proportion of mutations in portions of P. falciparum gene encoding kelch(K-13)-propeller domains (confering resistance to artemisinin)
incidence of adverse events | day 42
  monitoring of all adverse events experienced by participants

CONTACTS AND LOCATIONS:
Overall Officials: Gauthier Mesia Kahunu, PhD, Principal Investigator — University of Kinshasa
Locations (6):
- Democratic Republic of the Congo (6):
  - Centre Evangélique de Coopération, Kimpese, Bas-Congo Province
  - Centre de Santé Lupidi 1, Kapolowe, Haut-Katanga
  - Centre de Santé de Référence Mikalayi, Kazumba, Kasai-Central
  - Centre de Santé de Référence Rutshuru, Rutshuru, North Kivu
  - Centre de Santé Foyer Social, Kabondo, Tshopo
  - Centre de santé Bolenge, Bolenge, Équateur Province

IPD SHARING:
Plan to Share IPD: Undecided